CLINICAL TRIAL: NCT03987152
Title: Treatment of Congenital Vascular Malformations Using Sirolimus: Improving Quality of Life
Acronym: Sirolimus
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 57911; 2016-002157-38 (EudraCT Number)
Record Dates: First submitted 2019-03-01; First posted 2019-06-14 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2020-10

CONDITIONS: Vascular Malformations
Keywords: Sirolimus; mTor inhibitor; Quality of life; mammalian target of rapamycin (mTOR)
MeSH Terms: conditions — Vascular Malformations; Hereditary Sensory and Autonomic Neuropathies | interventions — Sirolimus

STUDY DESIGN:
Intervention Model Description: Challenge-Dechallenge-Rechallenge design All patients receive Sirolimus during challenge phase (6 months), stop Sirolimus during dechallenge phase (12 months), and if pain/symptoms returns Sirolimus intake is restarted during the rechallenge phase.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sirolimus (Other): Sirolimus administration: during Challenge and Rechallenge phase. Compared with the period 2 months before start of Sirolimus.
  Interventions: Drug: Sirolimus

INTERVENTIONS:
Drug: Sirolimus — Daily intake of Sirolimus during Challenge and Rechallenge phase
  Other Names: No other treatment

SUMMARY:
Congenital vascular anomalies are uncommon and belong to the group of rare diseases.These vascular malformations can cause serious complications including obstruction of vital organs and their function, recurrent infection and significantly reduced quality of life of persons affected.Treatment options range from conservative to surgical extirpation or intralesional embolisation/sclerosis. Unfortunately, this is often not enough. Many patients still have complaints like severe pain and invalidation due to the lymphatic or venous malformation making a normal functional life impossible. Recent case reports mention the positive effects of refractory patients with Sirolimus. Sirolimus, also known as rapamycin, is currently the only FDA-approved mammalian target of rapamycin (mTOR) inhibitor.

DETAILED DESCRIPTION:
Congenital vascular anomalies are uncommon and belong to the group of rare diseases. In 1996, the International Society of the Study of Vascular Anomalies adopted a new classification, distinguishing vascular malformations from vascular tumors. This classification was revised in 2014 and newly identified genetic features were taken into account. Vascular malformations feature dysplastic malformed vessels and are a consequence of a defective development of the embryonic vascular system. Vascular malformations can involve lymphatic vessels, capillaries, veins and arteries or even combinations. These vascular malformations are present at birth and grow with the child. Treatment options range from conservative to surgical extirpation or intralesional embolisation/sclerosis. Unfortunately, this is often not enough. Many patients still have complaints like severe pain and invalidation due to the lymphatic or venous malformation making a normal functional life impossible. These vascular malformations can cause serious complications including obstruction of vital organs and their function, recurrent infection and significantly reduced quality of life of persons affected. As the natural course of the disease affects multiple body systems, the therapeutic management is challenging. To date, no other medical treatment options are available. Although standard pain medication is given according the (inter) national pain protocols, patients still suffer pain and are not able to function normally in daily life. Majority (60-70% percent of the patients) of the patients is not able to have a normal life, with a normal job and normal social activities. Children are often not able to go to school normally, cannot play outside and have pain at the site of the malformation. The vast majority of literature reporting medical therapies for vascular anomalies consists of case reports and small series and is complicated by publication bias (negative findings are often not published), inconsistent use of nomenclature, and the absence of clinical trials. Recent case reports mention the positive effects of refractory patients with Sirolimus. Sirolimus, also known as rapamycin, is currently the only FDA-approved mammalian target of rapamycin (mTOR) inhibitor, indicated for prevention of kidney allograft rejection in adults and children 13 years or older, but is commonly used to manage organ rejection in younger children.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Congenital venous malformation, or lymphatic malformation or combined.
* Age older than 1 yr.
* Patients (or legal guardians for children) have to be able to sign the informed consent
* Patients are either refractory to standard care such as medical treatment (low molecular weight heparins, pain medication etc.), surgical resection and/or sclerotherapy/embolization (ineffective or accompanied by major complications) or there is no possibility for surgical intervention anymore. Only patients that have a normal clinical screening (no signs for infection, normal bone marrow function, normal liver and kidney function, normal glucose metabolism etc.) can be included.
* Patients included have no cardiac impairment
* Patients have no gastrointestinal impairment as Sirolimus is absorbed gastro-intestinal and normal function is needed
* No other underlying medical disorder like Down syndrome or other syndromes
* Women of reproductive age have to be informed that contraceptive methods are
* mandatory during the study time, pregnant women are excluded
* Karnofsky score > 50

Exclusion Criteria:

* No written informed consent
* Known hypersensitivity to drugs or metabolites from similar classes as study treatment.
* Patient has other concurrent severe and /or uncontrolled medical condition that would, in the investigator's judgment, contraindicated participation in the clinical study (e.g. acute or chronic pancreatitis, liver cirrhosis, active chronic hepatitis, severely impaired lung function with a spirometry ≤ 50% of the normal predicted value and/or O2 saturation ≤ 88% at rest, etc.)
* Recent history of primary malignancy ≤ 5 years
* Impaired cardiac function or clinically significant cardiac diseases
* Immunocompromised patients, including known seropositivity for HIV
* Patient with any other concurrent severe and /or uncontrolled medical condition that would,in the investigator's judgment, contraindicated participation in the clinical study.
* Pregnant or lactating women
* Karnofsky score < 50

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2017-09-18 (Actual); Primary Completion 2021-09-18 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
Quality of life using Sirolimus measured with survey (TAPQOL) | Change from baseline Quality of life at 6 months QoL in challenge phase, and 12 months QoL in Rechallenge phase.
  Quality of life: Questionnaire for Preschool Children's Health-Related Quality of Life (TAPQOL). Preschool Children Quality of Life, parent-reported questionnaire clustered into 12 multi-item scales, with higher scores range 0-100) indicating better HRQOL)
Quality of life using Sirolimus measured with survey (PedsQl) | Change from baseline Quality of life at 6 months QoL in challenge phase, and 12 months QoL in Rechallenge phase.
  Quality of life: Pediatric Quality of Life Inventory (PedsQl) (children) 23 items questionnaire, 0-100 scale, so that higher scores indicate better HRQOL (Health-Related Quality of Life). Psychosocial Health Summary Score, Physical Health Summary Score and Total score will be measured.
Quality of life using Sirolimus measured with survey (Research and development Rand-36). | hange from baseline Quality of life at 6 months QoL in challenge phase, and 12 months QoL in Rechallenge phase
  Quality of life: Rand-36 (adults) eight health domains; physical functioning, social functioning, role limitations due to physical health problems, role limitations due to emotional problems, mental health, vitality, pain and general health perception. Outcomes at each domain will be defined on a scale from a minimum score of 0 to a maximum score of 100. A higher score is equivalent to a better health.
Difference in pain scores after using Sirolimus measured with VAS score | Daily pain scores will be compared after 6 months in Challenge phase, after Challenge phase: starts the phase, and pain during 12 months in the Rechallenge phase
  Daily pain score (daily visual analogue scale (VAS-score 0-10) for children, and numeric rating scale (NRS-score 0-10) for adults)
Difference in pain scores after using Sirolimus measured with NRS score | Daily pain scores will be compared after 6 months in Challenge phase, after Challenge phase: starts the phase without Sirolimus treatment, and pain during 12 months in the Rechallenge phase
  Daily pain score (daily numeric rating scale (NRS-score 0 no pain -10 extreme pain) for adults)

SECONDARY OUTCOMES:
Return of pain after treatment and duration of lowered pain or pain free period in days | After 6 months Sirolimus intake till one year follow up.
  Amount of patients who have lowered pain or are pain free. Duration of lowered pain or pain free period in days.
Growth/progression of vascular malformation | MRI baseline compared with MRI after 6 months in challenge phase and 12 months in rechallenge phase
  MRI of the vascular malformation will be made at the beginning of the study and after six months of treatment with Sirolimus. An experienced radiologist will evaluate the evolution of the volume of the malformation.
Rate and occurence of adverse events related to Sirolimus | 4 years
  Adverse events: short and long term consequences of treatment with Sirolimus according to CTCAE version 5.0.
Severity of adverse events related to Sirolimus | 4 years
  Adverse events: short and long term consequences of treatment with Sirolimus according to CTCAE version 5.0.
Genetic mutations in the vascular malformation that can predict outcome of treatment with Sirolimus using Single Molecule Molecular Inversion Probes (smMIPs) | 4 years
  Secondary material that was obtained after surgery, stored in the HECOVAN biobank can be used for analyses. Comprehensive targeted Next Generation Sequencing screen using Unique Molecular Identifiers with a technical sensitivity of 1% mutant alleles was performed for frequently mutated positions using Single Molecule Molecular Inversion Probes. We will investigate if there is a correlation with a possible found mutation and painreduction or improvement of quality of life.
Pharmacogenetic profile in the vascular malformation that can predict outcome of treatment with Sirolimus | 4 years
  Genotyping will be performed using Taqman assays or Kompetitive Allele Specific PCR (KASPTM) assays in saliva swabs. Pharmacogenetic profiles (slow, intermediate, and extensive metabolizer) will be determined. Subjects compared on the outcome of sirolimus effectiveness for pain, and QoL stratified by CYP3A4.
Cost-effectiveness of administration of Sirolimus: Quality Adjusted Life Year (QALY) estimate for each patient | 4 years
  Via standardized questionnaires developed by the iMTA (institute for Medical Technology Assessment). The second part of the cost analysis consists of determining the cost prices for each volume of consumption.

CONTACTS AND LOCATIONS:
Overall Officials: Maroeska Loo, te, Dr., Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboudumc, HECOVAN workgroup, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Harbers VEM, Bouwman FCM, van Rijnsoever IMP, Verhoeven BH, van der Vleuten CJM, Schultze Kool LJ, de Laat PCJ, van der Horst CMAM, Kievit W, Te Loo DMWM. Magnitude and relevance of change in health-related quality of life in patients with vascular malformations treated with sirolimus. Front Med (Lausanne). 2023 Apr 20;10:1155476. doi: 10.3389/fmed.2023.1155476. eCollection 2023. PMID 37153086